CLINICAL TRIAL: NCT01394536
Title: The Effect of Overnight Use of Electroacustimulation on Postoperative Nausea and Vomiting in the Outpatient Surgery Population
Brief Title: Overnight Use of Electroacustimulation on Postoperative Nausea and Vomiting in the Outpatient Surgery Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed prior to enrollment of any subjects. No subjects were enrolled in this study.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-2010-0063
Record Dates: First submitted 2011-06-28; First posted 2011-07-14 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Post-operative Nausea and Vomiting
Keywords: Post-operative; post-op; nausea; vomiting
MeSH Terms: conditions — Vomiting; Nausea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Sham Comparator): "Sham" device - an EAS band placed over the P6 acupoint that will be turned off (inactive).
  Interventions: Device: Battery-operated electroacustimulation device (Inactive)
- 2 (Active Comparator): The second arm will use the ReliefBand (Aeromedix, Jackson, WY), an FDA-approved, reusable, battery-operated electroacustimulation device.
  Interventions: Device: Battery-operated electroacustimulation device (Active)

INTERVENTIONS:
Device: Battery-operated electroacustimulation device (Inactive) — In the sham arm, this device will not be turned on. The device to be used is the ReliefBand (Aeromedix, Jackson, Wy), an FDA-approved, reusable, battery-operated electroacustimulation device. The ReilefBand is a portable battery powered (lithium coin cells) device that is worn on the wrist like a watch. Two electrodes contact the skin with the aid of the application of electroconductive gel, and an electrical current of 25 mHz is transmitted through the skin. The device is applied at the Neiguan (P6) point, which is located on the inside of the wrist and is thought, in traditional Chinese medicine, to relieve nausea and vomiting (NV).
  Other Names: ReliefBand
  Arms: 1
Device: Battery-operated electroacustimulation device (Active) — The device to be used is the ReliefBand (Aeromedix, Jackson, Wy), an FDA-approved, reusable, battery-operated electroacustimulation device. The ReilefBand is a portable battery powered (lithium coin cells) device that is worn on the wrist like a watch. Two electrodes contact the skin with the aid of the application of electroconductive gel, and an electrical current of 25 mHz is transmitted through the skin. The device is applied at the Neiguan (P6) point, which is located on the inside of the wrist and is thought, in traditional Chinese medicine, to relieve nausea and vomiting (NV).
  Other Names: ReliefBand
  Arms: 2

SUMMARY:
Postoperative nausea and vomiting after outpatient surgery are significant sources of patient dissatisfaction. The prevention of postoperative nausea and vomiting (PONV) should be equally as important as prevention of pain because both are large sources of patient dissatisfaction and can necessitate admission after routine outpatient procedures.

None of the currently available pharmacological interventions are able to totally abolish PONV. The use of electroacustimulation is a useful adjunct in prevention of PONV, but has yet to be studied when the patient takes the device home with them after leaving an outpatient facility.

DETAILED DESCRIPTION:
The goal of this project is to perform a pilot study to determine if sending patients home with the electroacustimulation device will decrease their PONV and subsequently increase their overall satisfaction.

The primary outcome will be post-operative nausea and vomiting scores on a scale of 1-10 based on surveys which will be performed at 30m, 60m, 120m, and 24h post-op.

Secondary outcomes will be the amount of rescue nausea medications required by the patients, time to discharge, subjective pain assessment and the impact of their symptoms on the activities of daily living since being discharged from the surgery center based on survey, and amount of narcotic received.

This project would also aim to reduce the amount of time patients spend in recovery post-operatively, reduce hospital admissions secondary to persistent nausea and vomiting, and educate students and trainees about alternative methods of treating and preventing postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

• scheduled for outpatient surgery procedure under general anesthesia

Exclusion Criteria:

* pregnancy
* currently experiencing menstrual symptoms
* cardiac pacemaker
* previous experience with acupuncture therapy
* pharmacologic treatment for nausea or vomiting in the 24 hours prior to surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Measure of post-operative nausea and vomiting scores | 24 hours
  The primary outcome will be post-operative nausea and vomiting scores on a scale of 1-10 based on surveys which will be performed at 30m, 60m, 120m, and 24h post-op.

SECONDARY OUTCOMES:
Measure of amount of rescue nausea medications required | 24 hours
  The amount of rescue nausea medications required by the patients, time to discharge, subjective pain assessment and the impact of their symptoms on the activities of daily living since being discharged from the surgery center based on survey, and amount of narcotic received.
Amount of time spent in recovery post-operatively | 24 hours
  This project would also aim to reduce the amount of time patients spend in recovery post-operatively, reduce hospital admissions secondary to persistent nausea and vomiting, and educate students and trainees about alternative methods of treating and preventing postoperative nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Marcus, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States